CLINICAL TRIAL: NCT04440891
Title: Application of Transcranial Magnetic Stimulation Coupled With Virtual Reality for Slowing the Rate of Cognitive Decline in Patients With Alzheimer's Disease
Brief Title: Application of TMS Coupled With VR for Slowing the Rate of Cognitive Decline in Patients With Alzheimer's Disease
Acronym: TMS_AD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruitment due to Covid. 3 subjects consented but did not start any study procedures or participate in the study.
Sponsor: Ali Rezai (Other)
Responsible Party: Sponsor-Investigator, Ali Rezai, Director, West Virginia University
Organization: West Virginia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1904522298
Record Dates: First submitted 2020-05-22; First posted 2020-06-22 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- TMS-Stimulation with X-Torp task (Experimental): TMS with VR 1 experimental arm
  Interventions: Device: TMS stimulation with X-Torp task
- TMS-Stimulation with MindMotion Go (Experimental): TMS with VR 2 experimental arm
  Interventions: Device: TMS-Stimulation with MindMotion Go
- TMS-Sham with X-Torp task (Sham Comparator): TMS sham control with VR 1
  Interventions: Device: TMS-Sham with X-Torp task
- TMS-Sham with MindMotion Go (Sham Comparator): TMS sham control with sham VR 2
  Interventions: Device: TMS-Sham with MindMotion Go

INTERVENTIONS:
Device: TMS stimulation with X-Torp task — TMS-Stimulation with X-Torp task
  Arms: TMS-Stimulation with X-Torp task
Device: TMS-Stimulation with MindMotion Go — TMS-Stimulation with MindMotion Go
  Arms: TMS-Stimulation with MindMotion Go
Device: TMS-Sham with X-Torp task — TMS-Sham with X-Torp task
  Arms: TMS-Sham with X-Torp task
Device: TMS-Sham with MindMotion Go — TMS-Sham with MindMotion Go
  Arms: TMS-Sham with MindMotion Go

SUMMARY:
This is a randomized sham control study to evaluate how repetitive Transcranial Magnetic Stimulation (rTMS), interactive cognitive training, or the combination of rTMS and cognitive training reduce the cognitive decline of patients diagnosed with Alzheimer's disease

DETAILED DESCRIPTION:
Participants may be assigned to one of four experimental arms (1-TMS-Stimulation with X-Torp task, 2-TMS-Stimulation with MindMotion Go, 3-TMS-Sham with X-Torp task, 4-TMS-Sham with MindMotion Go.) The study will be conducted in two phases. During Phase 1, participants will be randomized between experimental conditions 1 and 4. Data will be analyzed upon completion of Phase1 and Phase 2 will commence only if there is efficacy in the TMS arm. During Phase2, participants will be randomized to arms 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

Male or Female between 50-85 years of age

* Able and willing to give informed consent
* Probable AD consistent with NIA/AA criteria
* Modified Hachinski Ischemia Scale (MHIS) score of <= 4
* Geriatric Depression Scale (GDS) score of <= 6
* Mini Mental State Exam (MMSE) score 18-26. The MMSE adjusted scoring instructions may be followed for screening patients as applicable.

Exclusion Criteria:

* Unstable medical conditions
* Visual impairments
* Mobility limitations
* Cognition-enhancing medication unless on a stable dosage for at least 3 months before the start of the trial.
* History of epilepsy or seizure disorder
* History of psychosis
* Current thoughts of suicidal ideation or self-harm as assessed by the Columbia-Suicide severity rating scale score
* Progressive neurological disorder or focal signs of abnormality on neurological exam as conducted by a neurologist (other than current diagnosis of AD)
* Tinnitus
* Metal implants (excluding dental fillings)
* Possible pregnancy
* Substance use disorder within the past six months
* Have other mental or physical conditions that are inappropriate for study participation at PI's or delegated sub investigator's discretion.
* Intake of one or a combination of the drugs that may due to their significant seizure threshold lowering potential

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Cognitive Performance | 6 months after completion study procedure
  Change in cognitive task performance over time using the total score on the Mini Mental State Examination (range 0-30)

SECONDARY OUTCOMES:
Brain MRI | 6 months after completion of study procedure compared to screening
  Change in brain structure and function over time
Memory Performance | 6 months after completion of study procedure compared to screening
  Total recall on the California Verbal Learning Test - short form (range 0-36)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Haut, PhD, Study Chair — Rockefeller Neuroscience Institute; Victor Finomore, PhD, Study Director — Rockefeller Neuroscience Institute
Locations (1):
- West Virginia University Rockefeller Neuroscience Institute, Morgantown, West Virginia, United States